CLINICAL TRIAL: NCT01448616
Title: Effect of Tenofovir on Genital HSV Shedding: a Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Effect of Tenofovir on Genital Herpes Simplex Virus (HSV) Shedding
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: CONRAD (Other); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Anna Wald, Professor, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 41250
Record Dates: First submitted 2011-09-14; First posted 2011-10-07 (Estimated); Results first posted 2016-01-12 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Herpes Simplex Type II
MeSH Terms: interventions — Tenofovir; Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Run-in Phase (No Intervention): Women will first participate in a run-in phase with twice daily swabbing.
- Study Drug Phase: TDF (Experimental): Participants will take tenofovir disoproxil fumarate (TDF) tablets and apply a placebo vaginal gel. Participants will begin treatment and swab the genital region twice daily for 5 more weeks. Study drugs will be administered once daily.
  Interventions: Drug: TDF; Drug: Placebo Vaginal Gel
- Study Drug Phase: Vaginal TFV Gel (Experimental): Participants will take oral placebo tablets and apply a tenofovir 1% (TFV) vaginal gel. Participants will begin treatment and swab the genital region twice daily for 5 more weeks. Study drugs will be administered once daily.
  Interventions: Drug: Vaginal TFV Gel; Drug: Placebo Tablets
- Study Drug Phase: Double Placebo (Placebo Comparator): Participants will take oral placebo tablets and apply a placebo vaginal gel. Participants will begin treatment and swab the genital region twice daily for 5 more weeks. Study drugs will be administered once daily.
  Interventions: Drug: Placebo Vaginal Gel; Drug: Placebo Tablets

INTERVENTIONS:
Drug: TDF — Oral tenofovir will be administered as tablets. TDF (Viread®) tablets contain 300 mg of tenofovir disoproxil fumarate, which is equivalent to 245 mg of tenofovir disoproxil. Study participants are instructed to take the one tablet, by mouth, once each day without regard to meals.
  Other Names: Tenofovir disoproxil fumarate (TDF) oral tablets
  Arms: Study Drug Phase: TDF
Drug: Placebo Vaginal Gel — Study participants are instructed to insert one dose (the entire contents of one applicator) of product into the vagina once each day. They are instructed to insert their gel as close to the same time each day as possible.
  The placebo gel (known as the 'universal' placebo gel) is formulated to minimize any possible effects - negative or positive - on study endpoints.
  Other Names: Placebo gel
  Arms: Study Drug Phase: Double Placebo; Study Drug Phase: TDF
Drug: Vaginal TFV Gel — Tenofovir 1% gel (w/w) is a gel formulation of tenofovir. Study participants are instructed to insert one dose (the entire contents of one applicator) of product into the vagina once each day. They are instructed to insert their gel as close to the same time each day as possible.
  Other Names: Tenofovir 1% Vaginal Gel
  Arms: Study Drug Phase: Vaginal TFV Gel
Drug: Placebo Tablets — TDF placebo tablets are film-coated and contain denatonium benzoate, a bittering agent, in addition to other inactive ingredients. Study participants are instructed to take the one tablet, by mouth, once each day without regard to meals.
  Other Names: Oral placebo
  Arms: Study Drug Phase: Double Placebo; Study Drug Phase: Vaginal TFV Gel

SUMMARY:
The investigators propose a randomized, double blind, placebo-controlled, cross-over trial to evaluate the effect of oral and topical (vaginal gel) tenofovir on genital herpes simplex virus (HSV) shedding among herpes simplex virus type-2 (HSV-2) seropositive, human immunodeficiency virus (HIV) seronegative women. The investigators hypothesize that tenofovir will reduce genital HSV shedding compared to placebo.

DETAILED DESCRIPTION:
The investigators propose a randomized, double-blind, placebo-controlled, cross-over study of 55 adult, healthy women who are HSV-2 seropositive and HIV-1 seronegative. Women will first participate in a run-in phase with twice daily swabbing. Following 4 weeks of swabbing, participants will be randomized 2:2:1 to one of three groups: 1) oral tenofovir and placebo gel, 2) oral placebo and tenofovir gel, or 3) oral placebo and placebo gel. Participants will begin treatment and swab the genital region twice daily for 5 more weeks. Study drug will be administered daily.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18-50
* HSV-2 seropositive by the University of Washington (UW) Western blot
* History of recurrent genital herpes, with more than 4 recurrences but less than 10 in the last year or, if currently on suppressive therapy, with more than 4 recurrences but less than 10 in the year prior to starting suppressive therapy
* HIV negative
* General good health
* Willing to not use antiviral therapy (other than the study drug) for the duration of the study
* Willing to obtain a swab from genital secretions twice daily for the duration of the study
* Willing to use effective birth control
* Able to provide written informed consent at screening and enrollment

Exclusion Criteria:

* HIV positive or at high risk for HIV acquisition (intravenous drug user or HIV+ sex partner)
* Hepatitis B (HepB) antigen (Ag) positive, or at high risk for HepB acquisition and not vaccinated
* Have a history of adverse reaction to tenofovir and/or adefovir
* Immunosuppressive medications, except for intranasal or topical (not high potency) steroids.
* Any kidney disease, or renal insufficiency, defined as serum creatinine >1.5 mg/dl. Participants with a prior history of a single episode of pyelonephritis will be eligible.
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 times upper limit of normal
* Pregnancy, as confirmed by a urine pregnancy test, planning to become pregnant during the course of the trial, or breast-feeding.
* Serious medical conditions or active infections
* Any other conditions that in the judgment of the investigator would preclude successful completion of the clinical trial.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2012-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Wald, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington Virology Research Clinic, Seattle, Washington, United States

REFERENCES:
- [Derived] Johnston C, Harrington R, Jain R, Schiffer J, Kiem HP, Woolfrey A. Safety and Efficacy of Combination Antiretroviral Therapy in Human Immunodeficiency Virus-Infected Adults Undergoing Autologous or Allogeneic Hematopoietic Cell Transplantation for Hematologic Malignancies. Biol Blood Marrow Transplant. 2016 Jan;22(1):149-56. doi: 10.1016/j.bbmt.2015.08.006. Epub 2015 Aug 8. PMID 26265463
- [Derived] Bender Ignacio RA, Perti T, Magaret AS, Rajagopal S, Stevens CE, Huang ML, Selke S, Johnston C, Marrazzo J, Wald A. Oral and Vaginal Tenofovir for Genital Herpes Simplex Virus Type 2 Shedding in Immunocompetent Women: A Double-Blind, Randomized, Cross-over Trial. J Infect Dis. 2015 Dec 15;212(12):1949-56. doi: 10.1093/infdis/jiv317. Epub 2015 Jun 4. PMID 26044291

RESULTS

PARTICIPANT FLOW:
Groups:
- Observational Group: All enrolled participants completed 28 days of twice-daily genital swabbing for HSV DNA. Only women completing >90% of requested swabs were randomized.
- Oral TDF + Vaginal Placebo Gel: Women received daily TDF tablets at 300mg + "universal" placebo gel for daily application
- Oral Placebo + Vaginal Tenofovir 1% Gel: Participants received a matching oral placebo to study product and 40mg of TFV gel both to be used daily
- Placebo Oral + Placebo Vaginal Gel: This group received the matching placebos to both study products
Period: Lead-In (Observational Phase)
Arm/Group | Observational Group | Oral TDF + Vaginal Placebo Gel | Oral Placebo + Vaginal Tenofovir 1% Gel | Placebo Oral + Placebo Vaginal Gel
Started | 73 | 0 (N/A during observational phase as participants randomized subsequently) | 0 (N/A during observational phase as participants randomized subsequently) | 0 (N/A during observational phase as participants randomized subsequently)
Completed | 64 (Participants who swabbed >90% completed this phase and were randomized to treatment 2:2:1.) | 0 (completed >90% of sample collection to qualify for randomization for next phase) | 0 | 0
Not Completed | 9 | 0 | 0 | 0
Not completed — Collected no genital swabs | 3 | 0 | 0 | 0
Not completed — Collected <90% of required swabs | 6 | 0 | 0 | 0
Period: Study Drug (Treatment Phase)
Arm/Group | Observational Group | Oral TDF + Vaginal Placebo Gel | Oral Placebo + Vaginal Tenofovir 1% Gel | Placebo Oral + Placebo Vaginal Gel
Started | 0 (All qualifying participants from this group moved to treatment group.) | 24 | 27 | 13
Completed | 0 | 22 | 23 | 9
Not Completed | 0 | 2 | 4 | 4
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Never initiated study drug | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Participants were randomized 2:2:1 to one of the 3 treatment arms after completing the lead-in phase
Groups:
- Oral TDF + Vaginal Placebo Gel: Participants randomized to receive 300mg Tenofovir Disaproxil Fumarate (TDF) 1 tab daily + the universal placebo vaginal gel (4ml) to be used daily.
- Oral Placebo + Vaginal TFV Gel: Participants randomized to receive matching oral placebo tab once daily + tenofovir (TFV) 1% vaginal gel (40mg in 4ml) to be used daily
- Oral Placebo + Vaginal Placebo Gel: Participants received matching oral tab and placebo gel both to be used daily
- Total: Total of all reporting groups
Arm/Group | Oral TDF + Vaginal Placebo Gel | Oral Placebo + Vaginal TFV Gel | Oral Placebo + Vaginal Placebo Gel | Total
Number analyzed (Participants) | 24 | 27 | 13 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 27 | 13 | 64
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 39.1 [20.8 to 50.8] | 36.7 [21.1 to 50.7] | 41.0 [19.2 to 48.7] | 37.3 [20.8 to 50.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 27 | 13 | 64
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 27 | 13 | 64

OUTCOME MEASURES:

1. Primary Outcome: HSV Shedding Rate in Those Receiving Oral TDF, Vaginal TFV, or Double Placebo
Description: The within-person changes in rate of HSV shedding during study drug administration (treatment phase) compared with the rate of HSV shedding during lead-in observation phase in the same participants. We evaluated only weeks 2-5 of HSV shedding during the treatment phase in comparison with the 4 weeks of the lead-in phase. We excluded the first week of samples from the treatment phase in order to allow for physiologic run-in of the treatment. This is analyzed separately for each treatment arm and not compared between arms.
Time Frame: Comparison of 4 weeks of treatment phase with 4 weeks of lead-in phase
Population: This is the intent-to-treat population (all randomized participants returning at least 1 swab in each phase of study)
Measure: Number (95% Confidence Interval); unit: percentage of swabs positive (%)
Groups:
- Oral TDF + Vaginal Placebo Gel: tenofovir disoproxil fumarate (TDF): Oral tenofovir will be administered as tablets. TDF (Viread®) tablets contain 300 mg of tenofovir disoproxil fumarate, which is equivalent to 245 mg of tenofovir disoproxil. Study participants are instructed to take the one tablet, by mouth, once each day without regard to meals.
  placebo gel: Study participants are instructed to insert one dose (the entire contents of one applicator) of product into the vagina once each day. They are instructed to insert their gel as close to the same time each day as possible.
  The placebo gel (known as the 'universal' placebo gel) is formulated to minimize any possible effects - negative or positive - on study endpoints.
- Oral Placebo + Vaginal TFV Gel: Tenofovir: Tenofovir 1% gel (w/w) is a gel formulation of tenofovir. Study participants are instructed to insert one dose (the entire contents of one applicator 40mg/4ml) of product into the vagina once each day. They are instructed to insert their gel as close to the same time each day as possible.
  placebo tablets: TDF placebo tablets are film-coated and contain denatonium benzoate, a bittering agent, in addition to other inactive ingredients. Study participants are instructed to take the one tablet, by mouth, once each day without regard to meals.
- Oral Placebo + Vaginal Placebo: placebo tablets: TDF placebo tablets are film-coated and contain denatonium benzoate, a bittering agent, in addition to other inactive ingredients. Study participants are instructed to take the one tablet, by mouth, once each day without regard to meals.
  placebo gel: Study participants are instructed to insert one dose (the entire contents of one applicator) of product into the vagina once each day. They are instructed to insert their gel as close to the same time each day as possible.
  The placebo gel (known as the 'universal' placebo gel) is formulated to minimize any possible effects - negative or positive - on study endpoints.
Arm/Group | Oral TDF + Vaginal Placebo Gel | Oral Placebo + Vaginal TFV Gel | Oral Placebo + Vaginal Placebo
Number analyzed (Participants) | 24 | 27 | 13
percentage of swabs positive (%)
  Lead-in Phase | 22.9 [20.6 to 25.2] | 13.8 [12.1 to 15.7] | 21.3 [18.4 to 24.5]
  Treatment Phase | 19.5 [17.4 to 21.8] | 12.0 [10.3 to 13.9] | 20.4 [17.0 to 24.1]
Statistical Analysis 1: Comparison: Oral TDF + Vaginal Placebo Gel; For intent to treat analysis, difference between lead-in and treatment phase (within arm comparison); Test type: Superiority or Other; p = 0.086, Poisson GLME — ITT; Risk Ratio (RR) = 0.86, 95% CI 2-sided [0.71 to 1.01]
Statistical Analysis 2: Comparison: Oral Placebo + Vaginal TFV Gel; For intent to treat analysis, difference between lead-in and treatment phase (within arm comparison); Test type: Superiority or Other; p = 0.54, Poisson GLME — For intent to treat analysis, difference between lead-in and treatment phase (within arm comparison); Risk Ratio (RR) = 0.94, 95% CI 2-sided [0.75 to 1.16]
Statistical Analysis 3: Comparison: Oral Placebo + Vaginal Placebo; For intent to treat analysis, difference between lead-in and treatment phase (within arm comparison); Test type: Superiority or Other; p = 0.47, Poisson GLME; Risk Ratio (RR) = 0.90, 95% CI 2-sided [0.67 to 1.22]

2. Secondary Outcome: Within-person Changes in Log-copy Numbers of HSV
Description: The within-person changes in mean log-copy numbers of HSV shed during treatment phase (oral TDF, vaginal TFV, or double placebo) compared with the lead-in (observation) phase in the same participants. Each treatment arm is analyzed separately without comparison between arms.
  We evaluated only weeks 2-5 of HSV shedding during the treatment phase in comparison with the 4 weeks of the lead-in phase. We excluded the first week of samples from the treatment phase in order to allow for physiologic run-in of the treatment.
Time Frame: Comparison of 4 weeks of treatment phase with 4 weeks of lead-in phase
Population: Analysis is within person changes such that the observational group contributed to analyses of those persons in each treatment randomization group
Measure: Mean (95% Confidence Interval); unit: log-copy number of HSV DNA shed
Arm/Group | Oral TDF + Vaginal Placebo Gel | Oral Placebo + Vaginal Tenofovir 1% Gel | Placebo Oral + Placebo Vaginal Gel
Number analyzed (Participants) | 24 | 27 | 13
log-copy number of HSV DNA shed
  Lead-in Phase | 4.02 [3.21 to 5.29] | 4.47 [2.92 to 6.24] | 3.71 [2.78 to 5.54]
  Treatment Phase | 4.11 [3.23 to 5.39] | 4.40 [3.37 to 5.13] | 4.22 [3.35 to 5.45]
Statistical Analysis 1: Comparison: Oral TDF + Vaginal Placebo Gel; Intent to treat analysis; Test type: Superiority or Other; p = 0.18, Linear Mixed Effects Model; Change in log copies = -0.16, 95% CI 2-sided [-0.40 to 0.07]
Statistical Analysis 2: Comparison: Oral Placebo + Vaginal Tenofovir 1% Gel; Intent to treat analysis; Test type: Superiority or Other; p = 0.008, Linear Mixed Effects Model; Change in log copies = -0.50, 95% CI 2-sided [-0.86 to -0.13]
Statistical Analysis 3: Comparison: Placebo Oral + Placebo Vaginal Gel; Intent to treat analysis; Test type: Superiority or Other; p = 0.45, Linear Mixed Effects Model; Change in log copies = 0.16, 95% CI 2-sided [-0.27 to 0.60]

3. Secondary Outcome: Genital Lesion Rate
Description: The within person change in proportion of days with lesions between the lead-in (observational) and study drug (treatment) phase for each arm separately. No between arm comparisons were performed. We include intent to treat with all randomized participants as well as per protocol (persons receiving study drug for at least 30 days with 90% or better reported compliance per returned product counts).
  We evaluated only weeks 2-5 of HSV shedding during the treatment phase in comparison with the 4 weeks of the lead-in phase. We excluded the first week of samples from the treatment phase in order to allow for physiologic run-in of the treatment.
Time Frame: Comparison of 4 weeks of treatment phase with 4 weeks of lead-in phase
Measure: Number (95% Confidence Interval); unit: percentage of days with lesions (%)
Groups:
- Oral Placebo + Vaginal Tenofovir 1% Gel: Participants received a matching oral placebo to study product and 40mg/4ml of TFV gel both to be used daily
Arm/Group | Oral TDF + Vaginal Placebo Gel | Oral Placebo + Vaginal Tenofovir 1% Gel | Placebo Oral + Placebo Vaginal Gel
Number analyzed (Participants) | 24 | 27 | 13
percentage of days with lesions (%)
  Lead-in Phase | 11.8 [9.5 to 14.5] | 8.7 [6.8 to 10.9] | 13.6 [10.3 to 17.5]
  Treatment Phase | 11.6 [9.3 to 13.3] | 7.1 [5.3 to 9.2] | 14.7 [10.7 to 19.6]
Statistical Analysis 1: Comparison: Oral TDF + Vaginal Placebo Gel; Intent to treat analysis; Test type: Superiority or Other; p = 0.90, Poisson GLME; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.70 to 1.37]
Statistical Analysis 2: Comparison: Oral Placebo + Vaginal Tenofovir 1% Gel; Intent to treat; Test type: Superiority; p = 0.25, Poisson GLM; Risk Ratio (RR) = 0.80, 95% CI 2-sided [0.54 to 1.18]
Statistical Analysis 3: Comparison: Placebo Oral + Placebo Vaginal Gel; Test type: Superiority; p = 0.82, Poisson GLM; Risk Ratio (RR) = 0.95, 95% CI 2-sided [0.57 to 1.57]

4. Secondary Outcome: Asymptomatic Shedding (Shedding on Days Without Genital Lesions)
Description: Within person changes in shedding on days without lesions between the lead-in (observational) phase and the study drug (treatment) phase. Each arm is evaluated separately and no inter arm comparisons are made.
  We evaluated only weeks 2-5 of HSV shedding during the treatment phase in comparison with the 4 weeks of the lead-in phase. We excluded the first week of samples from the treatment phase in order to allow for physiologic run-in of the treatment.
Time Frame: Comparison of 4 weeks of treatment phase with 4 weeks of lead-in phase
Population: All randomized participants are included in ITT analysis. Per protocol analysis includes persons receiving 30 or more days of study drug with >90% adherence as documented by returned product counts.
Measure: Number (95% Confidence Interval); unit: % days with asymptomatic shedding
Arm/Group | Oral TDF + Vaginal Placebo Gel | Oral Placebo + Vaginal Tenofovir 1% Gel | Placebo Oral + Placebo Vaginal Gel
Number analyzed (Participants) | 24 | 27 | 13
% days with asymptomatic shedding
  Lead-in Phase | 17.5 [15.4 to 19.9] | 7.6 [6.2 to 9.1] | 14.4 [11.7 to 17.4]
  Treatment Phase | 13.7 [11.8 to 15.8] | 8.2 [6.8 to 9.9] | 12.1 [9.2 to 15.5]
Statistical Analysis 1: Comparison: Oral TDF + Vaginal Placebo Gel; Intent to Treat; Test type: Superiority or Other; p = 0.010, Poisson GLME; Risk Ratio (RR) = 0.74, 95% CI 2-sided [0.59 to 0.92]
Statistical Analysis 2: Comparison: Oral Placebo + Vaginal Tenofovir 1% Gel; Test type: Superiority; p = 0.09, Poisson GLM; Risk Ratio (RR) = 1.30, 95% CI 2-sided [0.9 to 1.76]
Statistical Analysis 3: Comparison: Placebo Oral + Placebo Vaginal Gel; Intent to treat analysis; Test type: Superiority; p = 0.47, Poisson GLM; Risk Ratio (RR) = 0.90, 95% CI 2-sided [0.67 to 1.22]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected during the course of the lead-in phase (4 weeks) and the treatment (study drug) phase (5 weeks) and final AEs were recorded at a post-treatment follow up telephone visit 2 weeks after completing the study products.
Description: Unscheduled study visits were conducted as needed to evaluate potential adverse events.
  Adverse events were systematically collected in daily participant diaries and queried at each biweekly study visit.
Arm/Group | Observational Group | Oral TDF + Vaginal Placebo Gel | Oral Placebo + Vaginal Tenofovir 1% Gel | Placebo Oral + Placebo Vaginal Gel
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/24 | 0/27 | 0/13
Other Adverse Events (participants affected / at risk) | 11/73 | 12/24 | 11/27 | 3/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Observational Group (N=73) | Oral TDF + Vaginal Placebo Gel (N=24) | Oral Placebo + Vaginal Tenofovir 1% Gel (N=27) | Placebo Oral + Placebo Vaginal Gel (N=13)
Diarrhea (Gastrointestinal disorders) | 0 | 5 | 0 | 0
Headache (Nervous system disorders) | 0 | 3 | 4 | 0 — Including previously diagnosed migraine
Nausea (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Candida Intertrigo (Infections and infestations) | 0 | 0 | 0 | 1
Vulvovaginitis (Reproductive system and breast disorders) | 2 | 1 | 2 | 1
Vulvovaginal pruritis (Reproductive system and breast disorders) | 1 | 1 | 1 | 2
Vulvovaginal burning (Reproductive system and breast disorders) | 0 | 0 | 2 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Upper Respiratory Viral Illness (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 2 | 0

LIMITATIONS AND CAVEATS:
The study was not powered to detect differences in lesion rate; the study was appropriately powered to detect a 50% decrease in viral shedding only, and therefore may have been underpowered to detect significant findings for secondary outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No